CLINICAL TRIAL: NCT03202394
Title: A Phase IIa, Placebo Controlled, Multicenter Pilot Study to Evaluate the Safety and Efficacy of BIO-11006 Inhalation Solution in Patients With Acute Respiratory Distress Syndrome
Brief Title: Evaluation of Safety & Efficacy of BIO-11006 Inhalation Solution in Patients With ARDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarck Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIM-CL-005
Record Dates: First submitted 2017-06-20; First posted 2017-06-28 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: intubation; aerosol; sepsis; edema
MeSH Terms: conditions — Respiratory Distress Syndrome; Sepsis; Edema

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio to either BIO 11006 125 mg twice daily (intervention) plus standard of care ventilation or placebo BID plus standard of care ventilation. Patients randomized to receive BIO 11006 or placebo will start dosing at the time of ventilation and continue for up to 30 days or length of ventilation (if shorter).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active intervention (Active Comparator): Patients will be randomized in a 1:1 ratio to either aerosolized BIO-11006 (125mg in 3mL half normal saline) intervention twice daily plus ventilation for up to 28 days or placebo.
  Interventions: Drug: BIO-11006
- Placebo intervention (Placebo Comparator): Patients will be randomized in a 1:1 ratio to either aerosolized placebo (3mL half normal saline) intervention twice daily plus ventilation for up to 28 days or active drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIO-11006 — Intervention involves aerosolized delivery of either the active drug or placebo by the "Aeroneb Pro nebulizer".
  Arms: Active intervention
Drug: Placebo — Intervention involves aerosolized delivery of either the active drug or placebo by the "Aeroneb Pro nebulizer".
  Other Names: Half Normal saline
  Arms: Placebo intervention

SUMMARY:
This Phase IIa pilot study is a placebo controlled, multicenter study to evaluate safety and efficacy of aerosolized BIO-11006 Inhalation Solution in ARDS patients. The subjects will be randomized 1:1 to either BIO-11006 125 mg twice daily plus standard of care or placebo plus standard of care. The treatment will continue for up to 28 days. The study will enroll up to 40 adult ARDS patients in up to eight sites within USA.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled, parallel-group Phase IIa pilot study of aerosolized BIO 11006 in patients with sepsis-induced acute respiratory distress syndrome (ARDS). All patients enrolled in the study will be ventilated. To be eligible for enrollment, patients must be adults who have sepsis-induced ARDS within 48 hours prior to enrollment, require intubation, and exhibit bilateral infiltrates consistent with pulmonary edema on the frontal chest radiograph within 48 hours of enrollment. Patients will be randomized in a 1:1 ratio to either BIO-11006 125 mg twice daily (BID) plus standard of care ventilation or placebo (half normal saline [HNS]) BID plus standard of care ventilation. Patients randomized to receive BIO-11006 or placebo will start dosing at the time of ventilation and continue for up to 28 days or length of ventilation (if shorter). Patients in both groups will receive best available standard of care treatment, including low-volume mechanical ventilation as indicated by clinical judgment and patient response. The maximum duration of treatment will be 30 days.

The primary objective of this study is to evaluate the safety and efficacy of aerosolized BIO-11006 at a dose of 125 mg BID in ventilated patients who have ARDS. Safety is the primary endpoint in this study and will be monitored by adverse event reporting, oxygenation, mortality, vital signs, ventilator-free days, and ICU-free days.

This study will enroll up to 40 adult patients with ARDS induced by sepsis who first met the Berlin Criteria for ARDS within 48 hours of enrollment, and who require intubation and exhibit bilateral opacities consistent with pulmonary edema on frontal chest radiograph within 48 hours of enrollment.

BIO 11006 Inhalation Solution drug product is formulated at a dosage strength of 41.67 mg/mL (125 mg/3 mL) as an aqueous solution containing sodium chloride and is intended for aerosol administration by the "Aeroneb Pro®" nebulizer to patients randomized to active treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided (or relative has) written informed consent and authorization for use and disclosure of protected health information
2. Has a clinical diagnosis of sepsis or septic shock defined as:

   * Known or suspected infection
   * Systemic inflammatory response syndrome (SIRS), defined as meeting at least 2 of the following 3 criteria for a systemic inflammatory response:

     * White blood cell count >12,000 or <4,000 or >10% band forms
     * Body temperature >38°C (any route) or <36°C (by core temperatures only: indwelling catheter, esophageal, rectal)
     * Heart rate >90 beats/min or receiving medications that slow heart rate or pace rhythm
3. Enrollment must occur within 48 hours of first meeting ARDS criteria per the Berlin definition of ARDS (ARDS Task Force 2012) and no more than 72 hours from the initiation of mechanical ventilation. (The bilateral opacities, respiratory failure, and decreased P/F ratio must all be present within a 24 hour time period of one another.):

   * Lung injury of acute onset, within 1 week of an apparent clinical insult, with progression of respiratory symptoms
   * Bilateral opacities on chest imaging not fully explained by effusions, lobar/lung collapse, or nodules.
   * Respiratory failure not fully explained by cardiac failure or fluid overload. (Need objective assessment (e.g. echocardiography) to exclude hydrostatic edema if no risk factor present.)
   * Decreased arterial partial pressure of oxygen (PaO2)/ fraction of inspired oxygen (FIO2) ratio while on a minimum Positive End Expiratory Pressure (PEEP) of 5 cm water (H2O):

     * Moderate ARDS: 101 to 200 mmHg (≤ 26.6 kPa)
     * Severe ARDS: ≤ 100 mmHg (≤ 13.3 kPa)

Exclusion Criteria:

1. Age < 18 years or >75 years old
2. Greater than 48 hours since first meeting ARDS criteria per the Berlin definition of ARDS
3. Pregnant or breastfeeding (negative pregnancy test required prior to randomization for female patients of childbearing potential.)
4. Prisoner
5. Any other irreversible disease or condition for which 6 month mortality is estimated to be > 50%
6. Moderate to severe liver failure (Child Pugh Score > 12)
7. Severe chronic respiratory disease with a PaCO2 > 50 mmHg or the use of home oxygen
8. Patient, surrogate, or physician not committed to full support (exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest).
9. Major trauma in the prior 5 days
10. Lung transplant patient
11. No consent/inability to obtain consent
12. Moribund patient not expected to survive 24 hours
13. World Health Organization (WHO) Functional Class III or IV pulmonary hypertension
14. No intent/unwillingness to follow lung protective ventilation strategy or fluid management protocol
15. Currently receiving extracorporeal life support or high frequency oscillatory ventilation
16. Known hypersensitivity to BIO 11006
17. Burn victims >20% Total Body Surface Area (TBSA) or with known airway inhalation injury

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-08-05 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 28 days
  Assessment of frequency, type, severity, and duration of treatment-emergent Adverse Events (AE) daily during 28 day treatment period, including clinically significant laboratory abnormalities

SECONDARY OUTCOMES:
Incidence of mortality | End of treatment period (28 days) and end of follow up period (180 days)
  Mortality will be assessed daily during treatment for 28 days and at day 180 after enrollment.
Number of Intensive Care Unit (ICU)-free days | 28 days
  Number of days not in the ICU assessed daily during the 28 day treatment period.
Number of ventilator-free days | 28 days
  Number of days off the ventilator assessed daily during 28 day treatment
Change in oxygen saturation / fraction of inspired oxygen (S/F) ratio | 28 days
  Change in theS/F ratio assessed daily during the 28 day treatment period
Change in pro-inflammatory biomarkers from baseline to end of treatment | pretreatment and end of treatment period (28 days)
  ARDS associated biomarkers will be measured in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Brian Dickson, MD, Study Chair — Biomarck Pharmaceuticals
Locations (5):
- United States (5):
  - University of Chicago Medicine, Chicago, Illinois
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Div of Allergy, Pulmonary, Critical Care, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No